CLINICAL TRIAL: NCT04140474
Title: Evaluation of the Archimedes ™ System for Transparenchymatous Access to Pulmonary Nodules.
Acronym: SATAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion difficulties
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RI18_0030 (SATAN)
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Bronchoscopy; Lung Cancer; Solitary Pulmonary Nodule
Keywords: bronchoscopy; Lung Cancer; Solitary Pulmonary Nodule
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Archimedes procedure (Experimental): All included patients will receive anesthesia consultation, biological assessment and chest CT scan in thin sections. A surgical treatment will always be planned after presentation of the file in a meeting of multidisciplinary consultation of thoracic oncology. The Archimedes® procedure will be performed during a bronchoscopy under general anesthesia. Immediate monitoring consisted in a chest x-ray 1hour after the procedure.
  Interventions: Device: Archimedes procedure

INTERVENTIONS:
Device: Archimedes procedure — All patients will initially have a scanner necessary for planning by the Archimedes system of the tunneling path. each patient will then undergo a general anesthesia as for any bronchoscopy. Then start the Archimedes procedure itself to reach the SPN

SUMMARY:
The aim of this study protocol is to evaluate the feasibility of biopsies using the new system called Archimedes® in 12 patients with solitary pulmonary nodules (SPN) suspicious of malignancy not accessible through current bronchoscopy techniques.

DETAILED DESCRIPTION:
Due to the improvement of screening techniques, the detection of peripheral and isolated lesions is an increasingly frequent situation. However these SPN cause difficulties in obtaining a sample. Indeed, current endoscopic techniques remain insufficient in terms of performance. Moreover, computed tomography-guided percutaneous needle biopsy despite a very good sensitivity has many limitations related to the size of the lesions, the accessibility and important complications. The Archimedes® system is an improved version of LungPoint® and combines 3D reconstruction of chest images with intraoperative radioscopy. It uses a catheter to access through the bronchial wall the pulmonary parenchyma and navigate to the SPN. All included patients will receive anesthesia consultation, biological assessment and chest CT scan in thin sections. A surgical treatment will always be planned after presentation of the file in a meeting of multidisciplinary consultation of thoracic oncology. The Archimedes® procedure will be performed during a bronchoscopy under general anesthesia. Immediate monitoring consisted in a chest x-ray 1hour after the procedure. Patients' participation in the study will stop once they benefit from their thoracic surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years with a suspicious nodule of malignancy (primary lung tumor or metastasis of another solid tumor whose largest diameter is greater than or equal to 8 mm):
* Not associated with endobronchial tumor visible during inspection of tracheobronchial tree with soft bronchoscope
* Located in any part of the lung more than 10mm from the pleura
* For which surgical management (atypical resection, lobectomy, bilobectomy or pneumonectomy) is planned after presentation of the file at a multidisciplinary consultation meeting on thoracic oncology of the Investigating Hospital Center
* Patient able to understand the course of the study and giving informed consent
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Threatening cardiac arrhythmias defined by a rhythm disorder dating discovered less than a month ago
* Myocardial infarction less than one month old
* Hypercapnic respiratory decompensation less than one month old
* coagulopathy
* Thrombocytopenia with platelet count <100,000 / mm3
* Antecedent (ATCD) of significant bleeding during previous bronchoscopy
* ATCD of pulmonary arterial hypertension (PAH) or suspicion of PAH defined by a measurement of systolic pulmonary arterial pressure greater than 50 mmHg on echocardiography (this examination is not systematic but the suspicion of PAH on the thoracic CT scan leads to other cardiac echocardiographic examinations or right heart catheterization in case of inconclusive ultrasound)
* ATCD of pneumonectomy
* Giant bubble> 5cm located near the nodule or the tunneling path
* Inability to stop anticoagulant or antiplatelet therapy before the procedure (taking acetylsalicylic acid at any dose is allowed)
* Pregnant or lactating woman
* ATCD for thoracic radiotherapy on the nodule side
* Patient under tutorship or curatorship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Number of diagnostics obtained with the Archimedes system | Month 1
  It will be the biopsy yield defined as the number of patients in whom the results of nodule biopsies performed with the Archimedes® system are consistent with the surgical specimen.

SECONDARY OUTCOMES:
Scheduling time of the procedure | Day 21
  Procedure scheduling time defined by the number of minutes elapsed between recording the patient's chest scanner on the console and when the tunneling path was examined, selected, and exported
Access time to the nodule | Day 21
  Nodule access time defined as the number of minutes elapsed between the start of navigation and the placement of the sheath within the SPN
Fluoroscopy time | Day 21
  Fluoroscopy time defined by the number of minutes the patient is exposed to ionizing radiation
Patient registration time | Day 21
  Patient recording time defined as the number of minutes required to correlate the patient's position through fluoroscopy with the navigation aid system.
morbi-mortality | Month 1
  number of hemoptysis and pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Thomas EGENOD, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- CHU de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No